CLINICAL TRIAL: NCT02915809
Title: A Randomized, Double-Blind, Multicenter Study to Compare the Immunological Efficacy and Safety of GC3110B With GCFLU Quadrivalent Inj. Administered Intramuscularly in Healthy Adults
Brief Title: A Study to Evaluate Efficacy and Safety of GC3110B in Healthy Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3110B_P3
Record Dates: First submitted 2016-09-25; First posted 2016-09-27 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Influenza, Human
Keywords: Influenza Vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GC3110B Vaccine Group (Experimental): Participants randomized to receive a single dose of GC3110B vaccine (Biological: GC3110B vaccine).
  Interventions: Biological: GC3110B vaccine
- GCFLU Quadrivalent Inj. (Active Comparator): Participants randomized to receive a single dose of GCFLU Quadrivalent Inj. vaccine (Biological: GCFLU Quadrivalent Inj. vaccine).
  Interventions: Biological: GCFLU Quadrivalent Inj. vaccine

INTERVENTIONS:
Biological: GC3110B vaccine — 0.5mL, Intramuscular
  Other Names: GC3110B
  Arms: GC3110B Vaccine Group
Biological: GCFLU Quadrivalent Inj. vaccine — 0.5mL, Intramuscular
  Other Names: GCFLU Quadrivalent Inj.
  Arms: GCFLU Quadrivalent Inj.

SUMMARY:
The purpose of this study is to evaluate immunological efficacy and safety of GC3110B versus GCFLU Quadrivalent Inj. among healthy adults in 18 to 60 years of age.

DETAILED DESCRIPTION:
Adults 18 to 60 years of age will be randomly assigned in a 1:1 ratio to receive either GC3110B or GCFLU Quadrivalent Inj.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 60 years
* Informed consent form has been signed and dated
* Able to comply with the requirements of the study

Exclusion Criteria:

* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components
* Personal history of Guillain-Barré syndrome
* Subjects with severe chronic disease who are considered by investigator to be ineligible for the study
* Subjects who received a vaccination within 28 days before enrollment or who are scheduled for another vaccination during the study
* Immunocompromised subjects with immunodeficiency disease or subjects receiving immunosuppressive or immunomodulating therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 414 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer Ratios of Antibodies to the GC3110B or GCFLU Quadrivalent Inj. | Day 0 (Pre-Vaccination) and Day 21 (Post-Vaccination)
  Geometric mean titers of antibodies will be assessed using the hemagglutination inhibition (HI) assay.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Pre-Defined Seroconversion Before and Following Vaccination | Day 0 (Pre-Vaccination) and Day 21 (Post-Vaccination)
  Seroconversion is defined as either a pre-vaccination titer <1:10 and a post-vaccination titer ≥ 1: 40 or a pre-vaccination titer ≥ 1:10 and a ≥ 4-fold increase in post-vaccination titer 21 days after vaccination.
Percentage of Participants Achieving Pre-Defined Seroprotection Before and Following Vaccination | Day 0 (Pre-Vaccination) and Day 21 (Post-Vaccination)
  Antibodies will be assessed using the hemagglutination inhibition (HI) assay. Seroprotection is defined as a titer ≥1:40 at pre-vaccination and 21 days after vaccination.
Number and Percentage of Participants Reporting Solicited Adverse Events Following Vaccination | Day 0 to Day 6
Number and Percentage of Participants Reporting Unsolicited Adverse Events Following Vaccination | Day 0 to Day 21

IPD SHARING:
Plan to Share IPD: No